CLINICAL TRIAL: NCT06233851
Title: Prospective Paediatric Cohort Study of Biomarkers in the Early Management of Mild Traumatic Brain Injury and Prediction of Persistent Post-concussion Symptoms
Brief Title: BLOOD BIOMARKERS in PAEDIATRIC MTBI
Acronym: t-BIOMAP
Status: Completed | Type: Observational
Sponsor: Pediatric Clinical Research Platform (Other)
Responsible Party: Principal Investigator, Sergio MANZANO, professor, Pediatric Clinical Research Platform
Other Study IDs: 2020-01533
Record Dates: First submitted 2024-01-16; First posted 2024-01-31 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- mTBI patient: Children <16 years-old who suffered a head trauma in the last 24 hours with signs of mild traumatic brain injury
- control: Children <16 years-old who have a scheduled blood test for any reason

SUMMARY:
The goal of this observational study is to identify blood biomarkers that could help in the management of paediatric patients with mild TBI. The main questions it aims to answer are:

1. How can blood biomarkers reduce unnecessary CT scan and reduce the length of stay at the emergency department?
2. How can blood biomarker predict post-concussion symptoms?

Participants will have a blood sample taken when they are admitted at emergency department and will receive a questionnaire describing their symptoms 14 days and 3 months after their trauma.

DETAILED DESCRIPTION:
Mild Traumatic Brain Injury (mTBI) in children is a very frequent reason for presentation at the paediatric emergency department. In most cases, the trauma will not lead to intracranial lesions. The first objective for clinicians is therefore to detect all children in need of neurosurgical intervention after mTBI. Although computerized tomography (CT) is currently the modality of choice for acute intracranial haemorrhage identification, care should be taken to avoid unnecessary exposure to ionizing radiation in the developing brain. Monitoring the occurrence of bleeding usually involves an observation period which generally extends from six to twenty-four hours. This time is stressful for the child and parents as well as time and cost consuming for the hospital. In addition to the acute conditions, it has been described that post-concussion symptoms can occur in the weeks or months following the trauma, and neuropsychological follow-up of these children could help prevent or reduce the symptoms. The aim of our study is to find biomarkers that can identify children with clinically important intracranial injury and/or children that will eventually suffer from a post-concussion syndrome.

ELIGIBILITY:
Inclusion Criteria:

* mTBI within 24 hours

Exclusion Criteria:

* refusal of child or parents
* evidence of intoxication with alcohol or other substances
* history of TBI ( less than one month)
* epilepsy, encephalitis, meningitis, melanoma

Ages: 0 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: paediatric patient suffering from a mild TBI within 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
intracranial injuries on CT scan | Admission; within 24 hours
  Hemorrhage, oedema, traumatic infarction, diffuse axonal injury, pneumocephalus
Post concussion symptoms | 3 months
  Such as persistent headache, fatigue, concentration difficulty etc. Evaluated by a neuropsychologist and results of the PCSI score (post concussion symptoms inventory)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Manzano, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- HUG, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No